CLINICAL TRIAL: NCT01843543
Title: Assessing the Therapeutic Effect of Mindfulness-based Stress Reduction Intervention in Women With Urgency Incontinence Using Advanced Brain Imaging
Brief Title: Examining Bladder Control Using Mindful Based Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Rahel Nardos, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU_9405
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Urinary Urgency Incontinence
Keywords: Functional MRI (fMRI); Resting state functional connectivity MRI (rs-fcMRI); Diffusion Tensor Imaging (DTI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBSR participants (Experimental): Subjects in this arm will participate in an 8 week Mindfulness Based Stress Reduction Course
  Interventions: Other: Mindfulness Based Stress Reduction Course
- No MBSR Participants (No Intervention): Subjects in this arm will not participate in the Mindfulness Based Stress Reduction Course.

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction Course — The MBSR course developed by Jon Kabat-Zinn is a mind-body intervention that incorporates mindfulness techniques. This is an eight week MBSR course at OHSU. Class instruction will be augmented by daily home practices of listening to audiotapes, diary reflections, and reading preloaded on itouch devices provided to participants. Adherence will be assessed through in-house iMINDr tracking program loaded on the itouch.
  Arms: MBSR participants

SUMMARY:
Urgency Incontinence (where the bladder muscles contract suddenly, causing an immediate urge to urinate that is difficult to prevent) is commonly experienced in patients with overactive bladder. New findings have discovered that urgency incontinence may be connected to the interactions of certain regions of the brain and the bladder. Although this is a common problem, researched still do not know how these interactions impact the process of urgency incontinence. Furthermore, there is preliminary data to suggest that interventions such as Mindful-Based Stress Reduction (MBSR) can potentially be used as therapy for UI. The purpose of this study is to determine the impact MBSR training on UI symptoms, quality of life, and anxiety measures.

DETAILED DESCRIPTION:
Urgency Incontinence (where the bladder muscles contract suddenly, causing an immediate urge to urinate that is difficult to prevent) is commonly experienced in patients with overactive bladder. New findings have discovered that urgency incontinence may be connected to the interactions of certain regions of the brain and the bladder. Although this is a common problem, researched still do not know how these interactions impact the process of urgency incontinence. Furthermore, there is preliminary data to suggest that interventions such as Mindful-Based Stress Reduction (MBSR) can potentially be used as therapy for UI. The purpose of this study is to determine the impact MBSR training on UI symptoms, quality of life, and anxiety measures.

To determine the impact of MBSR training on Urinary Incontinence(UI) symptoms, quality of life and anxiety measures in women affected with UI. We hypothesize that participants will have significant improvement in UI and anxiety related symptoms and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with urinary urgency incontinence
* 40-85 years of age without a history of incontinence surgery
* current overactive bladder symptoms including urgency and urgency incontinence daily for the previous three months
* willing and able to complete all study related measures

Exclusion Criteria:

* medical contraindications for MRI scanning
* past or present overt neurological disease
* history of pelvic irradiation or bladder cancer
* current urinary tract infection
* current pelvic pain or painful bladder disorder
* symptomatic pelvic organ prolapse
* anticholinergic medication use within 2 weeks of baseline assessments
* past nonpharmacologic treatment for UI
* history of structured mindfulness based course or therapy

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Functional Magnetic Resonance Imaging (fMRI) | Administered before and within 6 weeks after participation in the MBSR course
  To use advanced brain imaging techniques, namely functional MRI (fMRI) to determine whether change in Urinary Incontinence and anxiety symptoms after a Mindfulness Based Stress Reduction course are associated with changes in activation patterns in the brain.

SECONDARY OUTCOMES:
Change in Overactive Bladder Symptom and Quality of Life Short Form | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  A questionnaire validated for overactive bladder patients that includes symptom bother and health-related quality-of-life questions
Change in Patient Global Impression of Severity and Improvement | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  single-question global indexes for Urinary Incontinence severity and improvement
Change in Beck Anxiety Inventory | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  A self-report questionnaire for anxiety consisting of 21 items with items describing physical, physiological and cognitive aspects of anxiety
Change in Mindfulness Attention Awareness Scale | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  A 15 item trait measure of the tendency to attend to present moment experiences in everyday activities
Change in Perceived Stress Scale | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  A 10 item self report questionnaire aimed to tap experiences of distress related to 'how unpredictable, uncontrollable, and overloaded respondents find their lives
Change in Urogenital Distress Inventory - Short Form | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  A 6 item self report questionnaire with items assessing life quality and symptom distress for urinary incontinence
Change in Urinary Incontinence Episodes in 3-Day Period | Administered before and within 6 weeks after participation in the MBSR course. Repeated between 6-8 months post intervention
  Subjects will be asked to keep a diary that tracks their bladder and urinary habits for 3 days
Change in Resting State Functional Connectivity Magnetic Resonance Imaging (rs-fcMRI) | Administered before and within 6 weeks after participation in the MBSR course
  To use advanced brain imaging techniques, namely functional connectivity MRI to determine whether change in Urinary Incontinence and anxiety symptoms after a Mindfulness Based Stress Reduction course are associated with changes functional connectivity patterns in the brain.
Change in Diffusion Tensor Imaging (DTI) | Administered before and within 6 weeks after participation in the MBSR course
  To use advanced brain imaging techniques, namely diffusion tensor Imaging(DTI) to assess white matter integrity and fiber tracking.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health Science University, Portland, Oregon, United States